CLINICAL TRIAL: NCT02161068
Title: Chart Review/PKD Genotyping
Brief Title: Clinical Care of Autosomal Polycystic Kidney Disease: Retrospective Analysis and Prospective PKD Genotyping
Acronym: ADPKD
Status: Completed | Type: Observational
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1308014251
Record Dates: First submitted 2014-04-23; First posted 2014-06-11 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: ADPKD
Keywords: ADPKD; Chart Review; PKD Genotyping
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — After informed consent is obtained, blood samples for PKD genotyping will be obtained from the study patient. Genotype results will be made available to the patient and they will be referred to a genetic counselor at their request. This service would not be a part of the study and therefore, genetic counseling would be done at the patient's expense.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective analysis to include demographic, clinical, biochemical, and genetic data that will further explore the natural history of ADPKD and assess the factors that are likely to be associated with the progression of disease and the incidence of complications including progressive chronic kidney disease, cardiovascular disease, and cerebrovascular disease.

DETAILED DESCRIPTION:
To explore questions regarding the natural history of PKD, as well as other, unforeseen issues, a comprehensive database of demographic, clinical, biochemical, and genetic data is required. This descriptive retrospective study can serve as a source of information regarding either the entire ADPKD population, or subsets of patients with specifically targeted characteristics. This will inform future prospective studies that will be designed to address issues regarding the natural history and complications of ADPKD.

The goal of this project is to collect data from a large population of patients with PKD. Based upon the estimated prevalence of PKD (1:500 and 1:1000 live births), it is estimated that there may be 10,000 PKD patients in the New York City area. This sample size far exceeds any database established thus far. As many as 40% of affected PKD patients are reportedly unaware of a family history of this disease, in part because many patients may go undiagnosed until they present with a medical complication (e.g., hypertension, kidney failure). Furthermore, this initiative will provide an opportunity to compare data from racially diverse populations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have a confirmed ADPKD diagnosis.

Exclusion Criteria:

* Unable to provide informed consent for PKD Genotyping.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled in this study will have the diagnosis of ADPKD
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Natural history of ADPKD | Up to 11 years
  Retrospective review to determine clinical, genetic, and radiographic characteristics that may influence the incidence of renal and extrarenal complications of ADPKD and prospective PKD genotyping if not previously performed.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Blumenfeld, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States